CLINICAL TRIAL: NCT05632718
Title: Searching for the Optimal Exercise Training Regimen for Reducing Obesity Relapse in Post Bariatric Surgery Patients With Insufficient Weight Loss - BariOPTIMIZE Randomized Parallel-arm Clinical Trial
Brief Title: Is Resistance Exercise More Effective Than Endurance in Reducing Obesity Relapse in Post-bariatric Surgery Patients
Acronym: BariOptimize
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); Research Centre in Physical Activity, Health and Leisure, Portugal (Unknown)
Responsible Party: Principal Investigator, Tiago Montanha, MsC Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIAFEL2022
Record Dates: First submitted 2022-11-20; First posted 2022-12-01 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Bariatric Surgery Patients
Keywords: Bariatric surgery; Resistance exercise; Resting metabolic rate
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single center 3-parallel-arm open-label randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance group (Experimental): 16 weeks of resistance exercise-training.
  Interventions: Other: Exercise
- Endurance group (Experimental): 16 weeks of endurance exercise-training.
  Interventions: Other: Exercise
- Control group (No Intervention): Does not enrole in exercise-training programme.

INTERVENTIONS:
Other: Exercise — Resistance and endurance supervised exercise-training. The training programme will last for 16 weeks. Training sessions will be held at Porto Faculty of Sports, 3 times per week with the duration of 1 hour.
  Arms: Endurance group; Resistance group

SUMMARY:
The goal of this clinical trial is to compare the effects of resistance exercise and endurance in post-bariatric surgery patients with insuficcient weight loss. The main question it aims to answer is:

* Is resistance exercise more effective than endurance exercise in preventing obesity relapse in post-bariatric surgery patients with insuficcient weight loss?
* Is resistance exercise more effective than endurance exercise in increasing resting metabolic rate in post-bariatric surgery patients with insuficcient weight loss?

Participants will be randomly assigned to one of the following groups:

* Resistance group: performing resistance exercise-training for 16 weeks
* Endurace group: performing endurance exercise-training for 16 weeks
* Control group: no intervention / standard medical care

DETAILED DESCRIPTION:
As lean body mass losses following bariatric surgery (BS) negatively affect resting metabolic rate (RMR), metabolic regulation and physical function, the researchers hypothesize that resistance exercise (REx) could more effectively prevent obesity relapse following BS. Also, the increased mechanical loading on lumbar spine intervertebral discs is associated with an ampered spinal health and low pressure pain threshold sensitvity in these patients. The main purpose of this project is to determine which exercise mode is best suited to prevent obesity and increase RMR of post-BS patients with insufficient weight loss.

To accomplish this, the researchers will perform a single center 3-parallel-arm open-label randomized clinical trial to determine if resistance exercise is superior to endurance exercise in reducing obesity relapse in post-BS patients with insufficient weight loss.

Aditionally we aim to investigate if resistance exercise is more effective than endurance exercise in producing changes in pressure pain threshold, spine mobility and thoracolumbar strength in post-BS patients with insufficient weight loss.

Patients will be enrolled in 4 (possibly 5) consecutive cohorts of n=20. These must be between 18 and 65 years old and have performed bariatric surgery in the prior 18 to 24 months. Participants will be randomly assigned one of three groups: control (CON), resistance exercise (REx) and endurance exercise (EEx), while the latter two will be enrolling exercise-training programs. All the groups will be assessed in two moments: baseline and 16 weeks (end of exercise programme). Both the training sessions and the assessments will be performed at Porto Faculty of Sports (FADEUP).

The study is expected to run for 2.5 years while including 5 cohorts of patients.

Participants will be the chance to participate for free in exercise sessions (REx, EEx ) and to have free access to the results of health evaluations performed. Main risks for participants in the study will be the potential adverse events associated with exercise or physical evaluations and the burden of time spent in exercise sessions and evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years (until the end of intervention)
* Having performed primary bariatric surgery (gastric sleeve or RYGB methods) in the prior 18 to 24 months in S. João Hospital center.
* Willing to participate and commit to intervention

Exclusion Criteria:

* Already taking part in a structured exercise programme.
* Presenting health condition contraindicating exercise practice
* Inability to commit with intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Percent fat mass | 16 weeks
  Change in fat mass percentage measured by DXA at 0 and 16 weeks (pre and post intervention)
Resting metabolic rate | 16 weeks
  Change in resting metabolic rate measured by indirect calorimetry at 0 and 16 weeks (pre and post intervention)

SECONDARY OUTCOMES:
Pressure Pain Threshold lumbar paraspinal | 16 weeks
  Change in Pressure Pain Threshold at 0 and 16 weeks (pre and post intervention)
Lean body mass | 16 weeks
  Change in lean body mass measured by DXA at 0 and 16 weeks (pre and post intervention)
Spine mobility, posture and stability | 16 weeks
  Change in spine mobility, posture and stability measured by algometer and Spinal Mouse and at 0 and 16 weeks (pre and post intervention)
Trunk muscle strength | 16 weeks
  Change in trunk muscle strength measured by dynamometry and expressed as peak torque relative to body weight at 0 and 16 weeks (pre and post intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- FADEUP, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No